CLINICAL TRIAL: NCT06649149
Title: The Effect of Gamified Instructional Material on Nursing Students' Therapeutic Communication Skills and Perception of Nursing Diagnoses in Aggressive Patient Management: A Randomized Controlled Trial
Brief Title: The Effect of Gamified Instructional Material on Nursing Students' Aggressive Patient Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Yadigar Ordu, Principal Investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Aggression Management
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: CONTROL; EXPERİMENTAL
Keywords: aggression; nursing students; game teaching; communication; nursing process
MeSH Terms: conditions — Aggression; Communication | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled trial in parallel groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Students will not know which group they are in. The data of the research will be entered by coding and the result evaluator will not know which group the students are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (Other): Students in the control group will be given a case discussion in a classroom environment.
  Interventions: Other: Education
- EXPERIMENTAL (Experimental): The students in the experimental group will play the game prepared for the case at https://genially.com/.
  Interventions: Other: Genially

INTERVENTIONS:
Other: Genially — In the study, an educational intervention will be prepared with the https://genially.com/ program, which is one of the interactive learning methods.
  Arms: EXPERIMENTAL
Other: Education — In the study, a case study prepared for the management of an aggressive individual will be discussed in a classroom environment.
  Arms: CONTROL

SUMMARY:
Purpose: This study aims to determine the effect of game-based learning on aggressive patient management of nursing students.

Material Method: The data of the study will be collected from senior nursing students in the 2024-2025 Academic Year using the "Participant Information Form, "Nursing Diagnosis Perception Scale" and "Therapeutic Communication Skills Scale for Nursing Students". The study is planned to be conducted in a randomized controlled trial design.

H.1. Subject: The effect of game-based learning on aggressive patient management of nursing students H.2. Purpose of the Study: This study aims to determine the effect of game-based learning on aggressive patient management of nursing students.

A case example for the management of an aggressive patient has been prepared by the researchers. The experimental group students will play the game prepared at https://genially.com/, which will be based on the prepared case. The control group students will handle the same case in class using the standard method.

Data will be collected using the "Participant Information Form", "Nursing Diagnosis Perception Scale" and "Therapeutic Communication Skills Scale for Nursing Students".

DETAILED DESCRIPTION:
Purpose: This study aims to determine the effect of game-based learning on aggressive patient management of nursing students.

Material Method: The data of the study will be collected from senior nursing students in the 2024-2025 Academic Year using the "Participant Information Form, "Nursing Diagnosis Perception Scale" and "Therapeutic Communication Skills Scale for Nursing Students". The study is planned to be conducted in a randomized controlled trial design.

H.1. Subject: The effect of game-based learning on aggressive patient management of nursing students H.2. Purpose of the Study: This study aims to determine the effect of game-based learning on aggressive patient management of nursing students.

A case example for the management of an aggressive patient has been prepared by the researchers. The experimental group students will play the game prepared at https://genially.com/, which will be based on the prepared case. The control group students will handle the same case in class using the standard method.

Data will be collected using the "Participant Information Form", "Nursing Diagnosis Perception Scale" and "Therapeutic Communication Skills Scale for Nursing Students".

The data of the study will be collected face-to-face with senior nursing students in the 2024-2025 Academic Year. Senior nursing students received theoretical training on the nursing process in the Fundamentals of Nursing course and on communication with specific groups in the Self-Awareness and Communication Methods course. The students also have clinical experience. Therefore, the study will be conducted with senior students. Within the scope of the study, the students will be given a theoretical training of a reminder nature by the responsible and assistant researcher on the nursing process and therapeutic communication. After the theoretical training, all randomly assigned class and play group students will be given the Participant Information Form, the Nursing Diagnosis Perception Scale and the Therapeutic Communication Skills Scale for Nursing Students and asked to fill it out (Pre-test). One week after the theoretical training, the students in the control group will process the cases and questions prepared by the researchers with the assistant researcher in class using question-answer, discussion and explanation methods. The cases and questions prepared by the researchers are given below. Expert opinions on the cases and questions are also obtained.

The case example that needs to be discussed in the classroom with the control group will be prepared as a game. https://genially.com/ will be used in the gamification of the case. Genially is a free platform that helps create interactive learning and communication materials with an easy-to-use content creation tool. Researchers have registered on this platform as instructors. They can create their own educational areas by using free content on this platform. With this method, the case example given above will be gamified with a GIF of an aggressive patient that can be accessed for free. Students will be presented with options and will be faced with guiding stimuli (such as "think again") in the answers they give incorrectly. Some questions in the game will be presented to students by dragging the answer options and placing them in the correct area. The prepared game link code will be created and sent to the students from the WhatsApp group that will be established. Students will be able to log in to the game by sharing the link. When the control group discusses the case, the experimental group will first be informed about the game and the link will be shared so that they can play the game. Then, students will be given the Nursing Diagnosis Perception Scale and the Therapeutic Communication Skills Scale for Nursing Students and asked to fill them out (Post-test). After the study is completed, the game link will be sent to all students in the control group and the other students in the class.

Data will be analyzed using the IBM SPSS 22 software package.

ELIGIBILITY:
Inclusion Criteria:

Having knowledge about the nursing process and therapeutic communication techniques

Exclusion Criteria:

Failure to participate in any research steps

Ages: 22 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Nursing Diagnosis Perception Scale (NDPS) | to two months
  Students' perception levels of nursing diagnoses will be determined.The maximum score that can be obtained from the scale is 5 points and the minimum score is 1. A low total score obtained from the scale indicates that nursing diagnoses are perceived positively.
Therapeutic Communication Skills Scale for Nursing Students (TCSSNS) | to two months
  Therapeutic communication skill levels of students will be determined. The highest score that can be obtained from the scale is 112, the lowest score is 16. An increase in the score obtained from the scale indicates an increase in therapeutic communication skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ordu Y, Aydin A. The effect of gamified teaching material on nursing students' therapeutic communication skills and perception of nursing diagnoses in aggressive patient management: A randomized controlled study. Nurse Educ Pract. 2025 Aug;87:104503. doi: 10.1016/j.nepr.2025.104503. Epub 2025 Aug 6. PMID 40784135